CLINICAL TRIAL: NCT07061158
Title: A Multidimensional Health Perspective: Analysis of the Effects of Yoga Intervention on Sleep Disorders in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yoga intervention
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Sleep Disorders; Insomnia; Aging; Yoga
Keywords: Yoga therapy; Older adults; Non-pharmacological intervention; Sleep quality; Multidimensional health; RCT
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Intervention Group (Experimental): Participants in this arm received a structured, age-appropriate yoga intervention for a period of 4 months. The program, delivered by certified yoga teachers, integrated physical postures, breathing exercises, and meditation/relaxation techniques designed to improve overall well-being.
  Interventions: Behavioral: Structured Yoga Course Intervention
- Usual Lifestyle Group (No Intervention): Participants in this arm maintained their usual lifestyle during the study period. They did not receive the yoga intervention from this study and only received routine health lifestyle guidance and follow-up. No form of exercise or psychological intervention was conducted during the study.

INTERVENTIONS:
Behavioral: Structured Yoga Course Intervention — Participants in this arm received a structured yoga course intervention for a period of 4 months. Sessions were held twice weekly, with each lasting 60 minutes. The curriculum was specifically designed to be gentle, slow-paced, and low-impact, making it suitable for older adults while emphasizing body awareness, mind-body integration, and psychological regulation. The course content included: breathing exercises (e.g., basic abdominal breathing combined with simple movements), asana (posture) practice (e.g., seated chair exercises, standing poses, prone poses, supine poses, and side-lying poses, emphasizing muscle activation, joint flexibility, body balance training, and coordination of breath with movement), and meditation and relaxation (e.g., supine rest, moon breath training, and OM chanting). All classes were instructed by experienced yoga teachers certified by the Yoga Alliance.
  Arms: Yoga Intervention Group

SUMMARY:
This randomized controlled trial aims to evaluate the impact of a structured yoga intervention on multidimensional health outcomes in older adults with sleep disturbances. A total of 62 participants aged 60 years and older with varying degrees of sleep disorders were recruited and randomly assigned to either a yoga intervention group or a control group. The intervention group received a standardized yoga program for 4 months, conducted twice weekly (60 minutes per session), and guided by certified instructors. The yoga intervention included physical postures, breathing exercises, and meditation/relaxation techniques. Health outcomes were assessed at baseline, mid-intervention (8 weeks), and post-intervention (16 weeks), across five domains: sleep quality, daytime functioning, cognitive performance, physical fitness, and emotional well-being. This study aims to explore the feasibility, safety, and integrative effects of yoga as a non-pharmacological intervention for promoting health in the aging population.

ELIGIBILITY:
Inclusion Criteria :

1. ≥ 60 years, conforming to the World Health Organization's definition of the elderly population.
2. Presence of varying degrees of sleep disorder symptoms (e.g., difficulty falling asleep, sleep maintenance difficulties, early morning awakening), but without severe mental illness or other significant underlying diseases affecting sleep (e.g., dementia, severe depression).
3. Possessing basic comprehension abilities, voluntarily participating in the study, and signing informed consent.
4. Capable of cooperating with follow-up and intervention.
5. No severe physical dysfunction, cardiopulmonary disease, or other conditions limiting participation in light physical activities (such as yoga practice).

Exclusion Criteria :

1. Severe mental disorders, such as schizophrenia, bipolar disorder, or severe depression.
2. Severe cognitive impairment, making it impossible to cooperate with the intervention and subjective questionnaire assessments.
3. Unstable cardiovascular diseases or other major organic diseases (e.g., recent myocardial infarction, end-stage renal failure).
4. Severe visual or auditory impairments that affect the safety and adherence to practice.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline, 2 Months Post-Intervention, and 4 Months Post-Intervention
  The Pittsburgh Sleep Quality Index (PSQI) is an internationally recognized self-rated questionnaire used to assess subjective sleep quality. A higher total score indicates poorer sleep quality. It encompasses seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. This study assesses changes in the PSQI total score to determine the impact of yoga intervention on the overall sleep status of older adults with sleep disorders.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | Baseline, 2 Months Post-Intervention, and 4 Months Post-Intervention
  The Epworth Sleepiness Scale (ESS) primarily assesses the likelihood of a participant experiencing sleepiness in various daily situations, serving as a common tool to measure daytime alertness. Higher scores indicate greater levels of sleepiness.
Fatigue Scale-14 (FSS-14) | Baseline, 2 Months Post-Intervention, and 4 Months Post-Intervention
  The Fatigue Scale-14 (FSS-14) assesses the subjective feeling of fatigue in daily life, reflecting the degree of exhaustion caused by sleep disorders. Higher scores indicate greater fatigue.
Montreal Cognitive Assessment-Beijing Version (MoCA-BJ) | Baseline, 2 Months Post-Intervention, and 4 Months Post-Intervention
  The Montreal Cognitive Assessment-Beijing Version (MoCA-BJ) is a widely used cognitive screening tool for older adults, covering multiple cognitive domains such as memory, attention, language, visuospatial ability, calculation, and orientation
Lower Limb Major Muscle Group Strength (Quadriceps Femoris, Hamstrings, Triceps Surae, Tibialis Anterior, Iliopsoas) | Baseline, 2 Months Post-Intervention, and 4 Months Post-Intervention
  Assesses the strength of major lower limb muscle groups, including the quadriceps femoris, hamstrings, triceps surae, tibialis anterior, and iliopsoas. Maximum isometric contraction values for both sides are recorded using a MICROFET2 standardized electronic dynamometer to comprehensively reflect individual lower limb support and gait stability.
Geriatric Depression Scale-15 (GDS-15) | Baseline, 2 Months Post-Intervention, and 4 Months Post-Intervention
  The Geriatric Depression Scale-15 (GDS-15) is suitable for rapid screening of depressive symptoms in older adults. Higher scores indicate a greater tendency towards depression.
Self-Rating Anxiety Scale (SAS) | Baseline, 2 Months Post-Intervention, and 4 Months Post-Intervention
  The Self-Rating Anxiety Scale (SAS) is used to assess subjective anxiety levels. Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sport University,, Beijing, Beijing Municipality, China